CLINICAL TRIAL: NCT01668238
Title: Detection of Benign and Malignant Thyroid and Breast Tumors by Fourier Transform Infrared Spectrometry
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: XU Zhi (Other)
Collaborators: Peking University (Other)
Responsible Party: Sponsor-Investigator, XU Zhi, Professor, Peking University
Organization: Peking University (Other)
Other Study IDs: PUCRP201105
Record Dates: First submitted 2012-08-07; First posted 2012-08-20 (Estimated); Last update posted 2012-08-20 (Estimated); Status verified 2012-08

CONDITIONS: Thyroid Tumor; Breast Tumor
Keywords: Thyroid tumor; Breast tumor; Fourier Transform Infrared Spectrometry; Tumor Diagnosis
MeSH Terms: conditions — Thyroid Neoplasms; Breast Neoplasms

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- malignant tumor: Inpatients with malignant tumors of thyroid and breast
- benign tumor: Inpatients with benign tumors of thyroid and breast
- Healthy volunteers: Volunteers without thyroid or breast tumors

SUMMARY:
The purpose of this stage of study is to establish discriminant among healthy tissue, benign and malignant thyroid and breast tumors by fourier transform infrared spectrometry variables.

DETAILED DESCRIPTION:
Recently,the methods to the diagnosis of tumors include palpation,X-ray,ultrasound,CT and MRI.The doctors could not get conclusion without a existing mass.The FNB is very popular nowadays in western countries,but it has been reported that about one-third malignant cases have been neglected by FNB,for the tissue isn't enough through the needle.There also have been reports about the increased auxilliary lymphnode metastases for breast cancer because of FNB.Although the Mammotome has been used widely,it is still traumatic.

Process of malignant transformation of tissues and cells, first proteins, lipids, carbohydrates and nucleic acids constitute the main substance of tissue and cell structure, conformation, and the number of occurrence of significant changes in subsequent histological changes. Fourier transform infrared spectroscopy is the major molecular bond coupling between the atoms vibrational spectra and molecular rotational spectra.

In this study, consists of three phases:

Stage one:

Continuous enrollment requires inpatient surgery 300 cases of thyroid cancer patients and breast cancer patients, 200 cases of preoperative determination of tumor on the surface infrared spectroscopy, infrared spectroscopy of the anterior tumor tissue and lymph node surgery, measured in vivo; at the same time into the group of 50 patients healthy people, the determination of surface infrared spectroscopy of the thyroid and breast area. Paraffin pathological findings as the gold standard, the thyroid and breast cancer patients were divided into the benign group and malignant group, relatively healthy and good, the distribution of differences of the surface infrared spectrum of malignant group, while relatively good in the malignant group IR spectra of the distribution of differences.

Phase II:

Were enrolled, infrared spectroscopy and pathological specimens were collected at different stages. Paraffin pathological findings as the gold standard, were established two tumor surface, the infrared spectra of the fresh in vitro and in vivo for tumor benign or malignant diagnosis discrimination system.

Phase III:

Into the infrared spectra collected data on behalf of the above-mentioned discrimination system to verify its sensitivity, specificity and accuracy; both paraffin pathological findings as the gold standard to compare the infrared spectral discrimination systems and intraoperative frozen section pathology for the diagnosis of benign and malignant tumors correctly rate differences, to explore the clinical value of infrared spectroscopy discrimination system.

ELIGIBILITY:
Patients:

1. Inclusion Criteria:

   * Patients undergoing thyroid and breast tumor surgery.
   * Informed consent form is signed.
   * An optical fibre and ATR probe can be applied to the operation field in process of open or laparoscopic surgery.
   * Male or female between the age of 18 to 80.
   * Patients can tolerate surgery and with non of these diseases: severe heart failure, liver failure, renal failure or respiratory failure.
2. Exclusion Criteria:

   * A state of emergency, such as Gastrointestinal bleeding, perforation, or acute obstruction.
   * unstable situation in operation, such as anesthetic accidents or intraoperative cerebral vascular accident.
   * From investigators' perspective patients do not suitable for the study

Healthy volunteers' inclusion criteria:

* Informed consent form is signed.
* No thyroid or breast cancer according to the professional judgment of general surgeon.
* No thyroid or breast disease according to thyroid function tests and breast type B-ultrasonic test within 3 months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Hospitalized patients undergoing thyroid and breast tumor sugery;
  2. Healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2011-08; Primary Completion 2012-09 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
pathologic findings | 12 months
  1. In operation patients, discriminant between benign and malignant thyroid and breast tumors are established by fourier transform infrared spectrometry variables, and pathologic diagnoses are gold standard.
  2. Between Patients and healthy volunteers, discriminant are established among thyroid and breast tumors and healthy tissues.

CONTACTS AND LOCATIONS:
Overall Officials: Zhi Xu, PhD MD, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China